CLINICAL TRIAL: NCT06503341
Title: Assessment and Control of Modifiable Risk Factors for Primary and Secondary Prevention
Brief Title: A Hospital-Based Registry of Preventive Cardiology Clinics
Acronym: PREVENT-CARD
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Dr Rubina Rauf, Assistant Professor Preventive Cardiology, National Institute of Cardiovascular Diseases, Pakistan
Other Study IDs: IRB-20/2023
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Morbidity; Cardiovascular Risk Assesment; Primary Prevention CVD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients: Adult patients with or without cardiovascular diseases.
  Interventions: Other: Cardiovascular risk assesment

INTERVENTIONS:
Other: Cardiovascular risk assesment — ASCVD Score and WHO Cardiovascular Risk score.

SUMMARY:
More research is needed to articulate the most effective ways to use these tools as screening tests in cardiovascular risk assessments and how they ultimately affect CVD mortality and morbidity outcomes. Clinicians are encouraged to continue sharing decision-making with patients to combine their unique cardiovascular risk factors and develop a comprehensive, effective treatment plan.

DETAILED DESCRIPTION:
Study Design: observational study Duration of Study: ongoing. Sample Size: All patients presenting to preventive cardiology clinics at the National Institute of Cardiovascular Diseases (NICVD), Karachi, Pakistan..

Sampling Technique: Non-probability consecutive sampling Data Collection Procedure: Verbal informed consent will be obtained from all the patients regarding their participation in the study and publication of study findings while maintaining confidentiality. Consecutive patients presenting preventive cardiology clinics at the National Institute of Cardiovascular Diseases (NICVD), Karachi, Pakistan, will be included in this registry. Demographic characteristics, physical examination, clinical history, risk modification, lab assessment, and ASCVD risk score at presentation and at every follow-up will be recorded using a structural questionnaire.

Data Analysis Procedure: The Tentative analysis plan uses collected data for research publications. The statistical package for social sciences (SPSS 21) will be used to analyze baseline characteristics. The Shapiro-Wilk test will be applied to check the hypothesis of normality for quantitative (continuous) variables. Descriptive statistics such as mean ± SD, median (IQR), skewness, maximum, and minimum will be calculated for quantitative (continuous) variables. Frequency and percentages will be calculated for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* All individuals attending the preventive cardiology clinics.

Exclusion Criteria:

* • Individuals who refused to give consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Both genders, age 18 and above, visiting preventive cardiology clinics with or without established CVD and may or may not have CVD risk factors.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2041-06 (Estimated)

PRIMARY OUTCOMES:
cardiovascular risk assesesment | Ten years
  risk stratification of Cardiovascular diseases (CVD) in patients without established CVD but with CVD co morbids.we are using Atherosclerotic Cardiovascular Diseases (ASCVD) Risk Score and World Heart Organization(WHO) Risk Score for CVD Risk Assesment. In ASCVD Risk Score, we categorize population into low risk ( score <5), borderline(score between 5 and 7.4) ,intermediate( score between 7.5 an 19.9) and high risk (score>20), using all parameters for risk assesment. For WHO risk score calculation we are using WHO Risk score system for South Asia. https://cdn.who.int/media/docs/default-source/cardiovascular-diseases/south-asia.pdf?sfvrsn=c5b0d9a3_2

SECONDARY OUTCOMES:
Cardiovascular risk reduction | Ten years
  CVD risk reduction in patients with or without established CVD but with CVD co morbids.
Cardiovascular related deaths | Ten years.
  Estimation of patients who expired in their follow up despite CVD risk factors management.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Rubina Rauf, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rauf R, Khan MN, Sial JA, Qamar N, Saghir T, Kazmi KA. Primary prevention of cardiovascular diseases among women in a South Asian population: a descriptive study of modifiable risk factors. BMJ Open. 2024 Nov 14;14(11):e089149. doi: 10.1136/bmjopen-2024-089149. PMID 39542488